CLINICAL TRIAL: NCT07334912
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicentre, Phase 2b Trial to Assess the Efficacy, Safety and Tolerability of AEF0217 for 24 Weeks in Adults and Older Adolescents With Down Syndrome.
Brief Title: AEF0217 in Participants With Down Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Collaborators: European Commission (Other); BioClever 2005 S.L. (Other); Eurofins ADME, S.L. (Unknown); Pharmalex (Unknown); Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEF0217-201; 2025-521013-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Down Syndrome (Trisomy 21)
Keywords: Down Syndrome; Trisomy 21; adaptative behaviour; cognitive impairments
MeSH Terms: conditions — Down Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: * Participants will be randomized in a 1:1:1:1 ratio to 1 of 4 groups to receive 1 of 3 doses of AEF0217 ( 0.1, 0.2 or 0.6 mg) or placebo
  * Randomization will be stratified by baseline IQ score 1) mild disability (IQ >55-70), 2) moderate disability (IQ >35-55] and by age group 3) older adolescent (≥16-<18 years) 4) adults (≥18 to ≤32 years)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor's team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AEF0217 0.1 mg (Experimental): 1 sachet of AEF0217 100µg + 1 sachet of Placebo
  Interventions: Drug: AEF0217 100 µg; Drug: Placebo
- AEF0217 0.2 mg (Experimental): 2 sachets of AEF0217 100µg
  Interventions: Drug: AEF0217 100 µg
- AEF0217 0.6 mg (Experimental): 2 sachets of AEF0217 300µg
  Interventions: Drug: AEF0217 300 µg
- Placebo (Placebo Comparator): 2 sachets of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AEF0217 100 µg — Sachet of granules
  Other Names: 3β-benzyloxy-17α-methyl-pregn-5-en-20-one
  Arms: AEF0217 0.1 mg; AEF0217 0.2 mg
Drug: AEF0217 300 µg — sachet of granules
  Other Names: 3β-benzyloxy-17α-methyl-pregn-5-en-20-one
  Arms: AEF0217 0.6 mg
Drug: Placebo — sachet of matching placebo granules
  Arms: AEF0217 0.1 mg; Placebo

SUMMARY:
The goal of this clinical trial is to identify if AEF0217 show an improvement in adaptive behaviors (daily life activities) in adults and older adolescents with Down Syndrome. It will also learn about the safety of AEF0217.

The main questions it aims to answer are:

* Does AEF0217 improve the daily life activities of the participants after being administered daily for 24 weeks ?
* Does AEF0217 improve fluid cognitive function (cognitive abilities that do not depend on prior knowledge) and the crystallised one (knowledge acquired through one's culture, including verbal ability and social knowledge), the quality of life and sleep of the participants after being administered daily for 24 weeks ?
* What medical problems do participants have when taking AEF0217?

Researchers will compare 3 doses of AEF0217 to a placebo (a look-alike substance that contains no drug) to see if AEF0217 improves adaptative behaviours in people with Down Syndrome.

Participants will:

* Take AEF0217 or a placebo every day for 24 weeks
* Visit the clinic 6 times with their caregiver for checkups, performing tests on a tablet and answering questionnaires.
* Be called by phone at home 5 times to check that they are well.

DETAILED DESCRIPTION:
This trial is a randomised, double blind, placebo controlled, parallel group, multicentre, Phase 2B trial.

Approximately 188 participants will be enrolled at clinical centres in Spain, France and Italy.

After the Day 1 visit (baseline) to the site and the Day 2 visit by phone/video, the trial will include 3 visits to the site during the treatment period, i.e., at the end of Weeks 4, 12, and 24, and there will be a follow-up visit 8 weeks after the end of treatment (in Week 32). Additional phone visits (via phone or video call) will be performed at the end of Weeks 1, 2, 8 and 18.

Participants completing 24 weeks of treatment will be invited to enter an open label 12-month extension trial (OLE) when it is approved and, if choosing to do so, will continue directly into the extension trial. . The participants who do not choose to enter the extension trial will enter the follow-up period. The participants that complete the trial, before the extension trial starts, may enter when it starts.

Safety assessments will be performed at each visit to the clinical site and include blood sampling for clinical chemistry, haematology and determination of AEF0217 and endocannabinoids concentrations at Weeks 12 and 24. In addition, urine samples will be collected.

Efficacy assessments will be performed during treatment at the end of Week 4 (adaptive behaviours, cognition and sleep efficiency), Week 12 (adaptive behaviours, cognition, quality of life, sleep efficiency and clinician functional assessment ), Week 24 (adaptive behaviours, cognition, quality of life, clinician functional assessment and sleep) and Week 32 at the end of the follow-up period (adaptive behaviours, cognition, sleep efficiency and clinician functional assessment) only for the participants who enter the follow-up period.

The total duration of the trial for an individual participant will be up to 36 weeks.

An independent (from the sponsor and the investigational centres) safety data monitoring committee (IDMC) will be set up in charge of performing an independent interim safety analysis at a minimum after 40 participants (at a minimum) have been treated for 12 weeks. The membership (including physicians with experience with Down syndrome and clinical pharmacologists), role and responsibilities of the IDMC will be defined in a specific charter before the trial starts. The IDMC will make recommendations related to any potential safety issues/signals to the Steering Committee of the trial (i.e., the coordinating investigator, the principal site investigator and responsible physician in each site and sponsor representatives

The trial will be conducted in accordance with the Declaration of Helsinki and ICH Good Clinical Practice.

Before initiating the trial, the clinical trial protocol, the written participant information and informed consent forms, the investigator's brochure, the recruitment material, and any other information for the participants and caregivers will be submitted to and approved by central ethic committees and national health authorities, as applicable.

Main Statistic analysis:

For the primary endpoint descriptive analysis will include: 1. The raw scores of the 9 subdomains of the VABS 3; 2. The raw scores of the 9 subdomains standardized to 100; and 3. Change from baseline to Week 24. These variables will be presented by treatment, dose, and visit (baseline and 24 weeks).

An MMRM will be used to evaluate the primary endpoint. The model will contain as dependent variable the change from baseline to Week 24 of the raw scores of the 9 subdomains of the VABS 3 standardized to 100 and as factors:

1. Treatment (placebo, AEF0217)
2. Dose (0 [placebo], 0.1, 0.2, 0.6 mg AEF0217) nested to treatment
3. Subdomains: receptive, expressive, written, personal, community, domestic, interpersonal relationships, play and leisure time, coping skills
4. Level of impairment at baseline
5. Treatment interactions with subdomain and/or level of impairment at baseline.
6. Dose interactions with subdomain and/or level of impairment at baseline

The model will use a restricted maximum likelihood (REML) method, and an unstructured covariance matrix will be used. If the model is not estimable, a compound symmetry structure will be used instead. The primary endpoint will be reached if there is a statistically significant (p<0.05) main effect of treatment or dose or any significant (p<0.05) interactions between treatment or dose and subdomain and/or the previous factors with the impairment at baseline.

For the other efficacy endpoints (secondary and exploratory) and pharmacodynamic endpoints the same model with the appropriate adaptations will be used as will be described in the SAP.

Safety endpoints: TEAEs will be reported in individual data listings and frequency tables. Based on reported terms, TEAEs will be coded in and tabulated by MedDRA SOC and PT. AEs will be classified based on severity (mild, moderate, severe) and causality (related or not related) and outcome.

Summary statistics of vital signs, ECG, and safety laboratory parameters (with flagging of values outside the normal ranges and considered clinically significant) will be provided.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female. For males: Throughout the trial and until the end of the trial, male participants should refrain from donating sperm and, if sexually active, use double-barrier contraceptive methods (i.e., male condoms and spermicide), or the female partner must use the same highly effective contraceptive methods as female trial participants .

For females: Female participants of childbearing potential, defined as having a menstrual cycle that is confirmed prior to enrolment, must use highly effective contraception throughout the trial and until 3 months after the last dose of the trial intervention, be sexually abstinent, or have a vasectomized partner.

* 2. Age ≥16 to ≤32years.
* 3. BMI ≥18.0 and ≤35 kg/m2.
* 4. Clinical diagnosis of Down syndrome (full trisomy 21 or translocations) documented by chromosomal analysis (karyotyping).
* 5. Must be independently mobile and have sufficient vision and hearing to participate in the trial evaluations.
* 6. IQ >35-70 measured with Leiter-3. Individuals with IQ from >35 to <40 must have adequate cognitive and behavioural abilities according to the judgment of the principal investigator.
* 7. VCI of WISC-V language test score >4, based on mental age (estimated via IQ).
* 8.Must be able to understand most of the time and to express if he/she does not understand to the extent that he/she can accept the trial procedures. Must not use other forms of communication, signs, symbol boards, or devices as his/her primary form of communication.
* 9. Must have a parent or other reliable caregiver who agrees to accompany the participant to all clinic visits, provide information about the participant as required by the protocol, and ensure compliance with the medication schedule and protocol requirements
* 10.The parent or caregiver must be a constant and reliable informant with sufficient contact with the participant to have detailed knowledge of the participant's adaptive functioning to be able to answer accurately the questions asked by a neuropsychologist at the assessments.
* 11. Vital signs, ECG , and safety laboratory3 parameters must be without clinically relevant abnormalities as per the judgement of the investigator, except for:

  * Stable type 1 or 2 diabetes provided the participant is monitored regularly prior to and during the trial to ensure adequate glucose control.
  * Hypothyroidism controlled by treatment so that the participant is euthyroid and T4 stable (range 77-155 nmol/L) for at least 6 weeks prior to randomization. Fluctuations in TSH up to a maximum of 10 mIU/L are allowed.
* 12. a. Assent by the participant and consent by the legally authorized representative(s) on behalf of the participant or b. Consent by the participant in situations where consent rather than assent can be provided by the participant.
* 13. Informed consent by the participant's caregiver to take on the obligations of the caregiver in this trial.

Exclusion Criteria:

* 1. Pregnant or nursing female. Down syndrome
* 2. Mosaic Down syndrome or Down Syndrome Regression Disorder (DSRD). Medical history and clinical status
* 3. Active or clinically relevant conditions that could, in the investigator's judgment, affect absorption, distribution, or metabolism of the trial medication (e.g., inflammatory bowel disease, gastric or duodenal ulcers or severe lactose intolerance); controlled celiac disease is allowed.
* 4. Clinically relevant obstructive pulmonary disease or asthma that is untreated. Patients well-controlled by treatment (inhalation or oral) for at least 6 weeks prior to screening may be included if considered safe by the investigator.
* 5. Known severe obstructive sleep apnoea or if the investigator thinks that the person should be referred for a diagnosis/treatment of obstructive sleep apnoea.
* 6. Recent (≤1 year) or ongoing haematologic or oncologic disorders (mild anaemia is allowed).
* 7. History of infantile spasms/convulsions/epilepsy, severe head trauma or central nervous system infections (e.g., meningitis), except for isolated events of febrile seizures more than 8 years ago.
* 8. Clinically relevant unstable gastrointestinal, renal, hepatic, endocrine (including metabolic syndrome), or cardiovascular system disease as per the investigator's judgement.
* 9. Any prevailing psychiatric disorder diagnosed using the DSM-5 that dominates a person's overall clinical condition outside of Down syndrome. If symptoms consistent with a diagnosis of psychiatric illness are detected during the screening assessment (NPI-Q) and considered as dominating, the investigator may request a psychiatric evaluation. If necessary, a consultant psychiatrist will be responsible for the final diagnosis, as this is not the investigator's responsibility.
* 10. Participants with secondary psychiatric disorders including conduct disorders, attention deficit hyperactivity disorder, depressive disorders, anxiety disorders, and others that: 1) dominate the overall clinical condition according to the investigator's assessment; and/or 2) are not stabilized by medical or behavioural treatments, a stabilized treatment being defined as a stable therapeutic regimen and dose for the 3 months prior to randomization; and/or 3) the type of pharmacological treatment is on the list of drugs that are prohibited.
* 11. Symptoms of early dementia confirmed by the NTG-EDSD.
* 12. Substance use disorder as defined by the DSM-5.
* 13. Positive urine test for alcohol and drugs of abuse at screening and prior to first dosing.
* 14. Current diagnosis of epilepsy.
* 15. A history of intentional self-harm or suicide attempts brought on by suicidal thoughts. Suicidal ideation in the 12 months before screening, even if there was no suicide attempt or intentional self-harm. Assessed using 3 distinct questions about suicidal behaviour, suicidal ideation, and any self-harming actions.
* 16. Known hypersensitivity to AEF0217 or fructose intolerance.
* 17. Clinically significant illness, such as active infections, within 2 weeks prior to randomization, according to the investigator's judgment.
* 18. Any current life-threatening disease.
* 19. Any additional clinically significant concomitant disease, condition, or screening result that, in the investigator's opinion, could endanger the participant's safety, interfere with trial conduct and related procedures, or influence how the trial results are interpreted.
* 20. Treatment with 1st generation neuroleptic drugs currently or within 3 months prior to randomization and benzodiazepines currently or in the 4 weeks prior to baseline assessments.
* 21. Intake of products containing EGCG (e.g., TEAVIGO, Mega Green Tea Capsules Life Extension, or Font-UP Grand Fontaine Laboratories) currently or during the last 4 weeks prior to the baseline assessments.
* 22. Treatment with medications or very regular consumption of fruits (i.e., pomelo/grapefruit) or natural remedies (i.e., hypericum preparations) known to strongly or moderately induce or inhibit CYP3A4/5 P450 isozymes..
* 23. Administration of an investigational medicinal product, including AEF0217, within the last 3 months prior to randomization.

Ages: 16 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the normalized scores of the 9 subdomains of the VABS-3 at week 24 (end of treatment) | Baseline and Week 24
  Raw scores will be normalised to 100. Higher scores on the VABS-3 indicate better adaptive functioning.

SECONDARY OUTCOMES:
Changes from baseline in the fluid cognition composite change sensitive score of the NIH-ToolBox for Intellectual Deficiencies at Week 24 (end of treatment) | Baseline and Week 24
  Higher scores on the NIH-TCB for ID indicate better performance
Changes from baseline in the individual change sensitive scores of the Flanker inhibitory control & attention test used to measure fluid cognition in the NIH-TB for ID at week 24 (End of treatment). | Baseline and Week 24
  Higher scores indicate better performance
Changes from baseline in the individual change sensitive scores of the Picture Sequence Memory test used to measure fluid cognition in the NIH-TB for ID at week 24 (End of treatment). | Baseline and Week 24
  Higher scores indicate better performance
Changes from baseline in the individual change sensitive scores of the List Sorting Working Memory test used to measure fluid cognition in the NIH-TB for ID at week 24 (End of treatment). | Baseline and Week 24
  Higher scores indicate better performance
Changes from baseline in the individual change sensitive scores of the Dimensional Change Card Sort test used to measure fluid cognition in the NIH-TB for ID at week 24 (End of treatment). | Baseline and Week 24
  Higher scores indicate better performance
Changes from baseline in the individual change sensitive scores of the Pattern Comparison Process Speed test used to measure fluid cognition in the NIH-TB for ID at week 24 (End of treatment). | Baseline and Week 24
  Higher scores indicate better performance
Changes from screening values used as baseline of the Verbal comprehensive Index of the WISC-V at Week 24 (end of treatment). | Baseline and Week 24
  Higher scores on the VCI indicate better crystallized cognition
Changes from screening values used as baseline of the Vocabulary test of the WISC-V at Week 24 (end of treatment). | Baseline and Week 24
  Higher scores indicate better performance
Changes from screening values used as baseline of the "Similarities" test of the WISC-V at Week 24 (end of treatment). | Baseline and Week 24
  Higher scores indicate better performance
Changes from baseline of the total score of Generic Score Scale of the Peds-QL at week 24 (end of treatment) | Baseline and week 24
  Higher scores indicate better health-related quality of life
Changes from baseline t of the total score of the cognitive functioning scale of the Peds-QL at Week 24 (end of treatment) | Baseline and week 24
  Higher scores indicate better health-related quality of life
Changes from baseline of the total score of the Family Impact scale of the Peds-QL at Week 24 (end of treatment) | Baseline and week 24
  Higher scores indicate better health-related quality of life
Changes from baseline of the Psychosocial Health summary score of the of the Peds-QL at week 24 (end of treatment) | Baseline and week 24
  Higher scores indicate better health-related quality of life
Changes from baseline of the Physical Health summary score of the of the Peds-QL at week 24 (end of treatment) | Baseline and Week 24
  Higher scores indicate better health-related quality of life
Changes from baseline of the Parent HRQL summary score of the of the Peds-QL at week 24 (end of treatment) | Baseline and week 24
  Higher scores indicate better health-related quality of life
Changes from baseline of the Family Functioning summary score of the of the Peds-QL at week 24 (end of treatment) | Baseline and week 24
  Higher scores indicate better health-related quality of life
Changes from baseline of each mean scale scores of the domains composing the Generic Core Scale at Week 24 (end of treatment) | Baseline and week 24
  Mean scale scores will be analysed after normalisation to 100. Higher scores indicate better health-related quality of life
Changes from baseline of each mean scale scores of the domains composing the Impact Family Questionnaire at Week 24 (end of treatment) | Baseline and week 24
  Mean scale scores will be analysed after normalisation to 100. Higher scores indicate better health-related quality of life
Changes from baseline of the sleep efficiency score of the PSQI at Week 24 (end of treatment) | Baseline and week 24
  Lower scores indicate better sleep quality
Number of participants reporting a Treatment Emergent Adverse Event. | From Day 1 to Week 24 or Week 32
  Presented by treatment group ; End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
Percentage of participants with an Adverse Event | From Day 1 to week 24 or week 32
  Presented by treatment group ; End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
Number of events reported (AEs and TEAEs) | From Day 1 to week 24 or week 32
  Presented by treatment group ; End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
Incidence of treatment-related and not related TEAEs | From Day 1 to end of trial at week 24 or at week 32
  Compared by treatment group ; End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
Incidence of related or not Treatment Emergent SAEs | From Day 1 to week 24 or week 32
  Presented by treatment group ; End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
Vital Signs: Systolic Blood Pressure | Baseline and at week 4, week 12, week 24, week 32
  Changes in Systolic Blood Pressure (mmHg) over the study period
Vital Signs : Diastolic Blood Pressure | Baseline and at week 4, week 12, week 24, week 32
  Changes in Diastolic BP (mmHg) over the study period
Vital Signs : Heart Rate | Baseline and at week 4, week 12, week 24, week 32
  Changes in Heart Rate (bpm) over the study period
12 Lead ElectroCardiogram test | Baseline and at week 4, week 12, week 24, week 32
  Changes in 12-lead electrocardiogram (ECG) parameters in PR, QRS, QT, QTcF, and RR intervals over the study period
Changes from baseline in the total score of the Anxiety, Depression, and Mood Scale (ADAMS) at week 24 | Baseline and at week 24
  ADAMS questionnaire measures anxiety, depression and mood. Will be presented by treatment group.
  Range is 0 to 87 where higher scores are being indicative of more severe symptomatology.
Changes from baseline in the total score of the Anxiety, Depression, and Mood Scale (ADAMS) at week 32. | Baseline and at week 32
  ADAMS questionnaire measures anxiety, depression and mood. Will eb presented by treatment group. Range is 0 to 87 where higher scores are being indicative of more severe symptomatology.
Changes from baseline to the end of trial in the score of the manic/hyperactive behaviour subscale of the Anxiety, Depression, and Mood Scale (ADAMS) at the end of trial. | Baseline and at week 24 or at week 32
  End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
  Range is 0 to 15 where higher scores are being indicative of more severe symptomatology.
Changes from baseline in the score of compulsive behaviour subscale of the Anxiety, Depression and Mood Scale (ADAMS) at the end of trial. | Baseline and at week 24 or at week 32
  End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
  Range is 0 to 9 where higher scores are being indicative of more severe symptomatology.
Changes from baseline in the scores of the general anxiety subscale of the Anxiety, Depression and Mood scale (ADAMS) to the end of trial. | Baseline and at week 24 or at week 32
  End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
  Range is 0 to 21 where higher scores are being indicative of more severe symptomatology.
Changes from baseline in the scores of the depressed mood subscale of the Anxiety, Depression and Mood scale (ADAMS) to the end of trial. | Baseline and at week 24 or at week 32
  - End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
  Range is 0 to 21 where higher scores are being indicative of more severe symptomatology.
Changes from baseline in the scores of the social avoidance subscale of the Anxiety, Depression and Mood Scale (ADAMS) to the end of trial. | Baseline and at week 24 or at week 32
  End of trial is defined as week 24 if the participant enters in the open label extension trial or week 32 (end of follow-up) if not.
  Range is 0 to 21 where higher scores are being indicative of more severe symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Pier Vincenzo PIAZZA, MD, PhD, Study Chair — Aelis Farma; Rafael DE LA TORRE FORNELL, PharmD, PhD, Principal Investigator — Hospital del Mar Research Institute
Locations (10):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - Genetics department, Hospices Civils de Lyon, Lyon
  - Service Génétique Médicale, CHU de Montpellier, Montpellier
  - Genetics department, Institut Jérôme Lejeune, Paris
  - Service de Génétique, Chromosomique et Moléculaire, Chu de Saint Etienne, Saint-Etienne
- Italy (3):
  - IRCCS Istituto Delle Scienze Neurologiche, Azienda Unita Sanitaria Locale Di Bologna, Bologna
  - Centro di Medicina dell'Invecchiamento, Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - UOR of Neurofarmacology and Translational Neurosciences, Associazione Oasi Maria S.S.Onlus, Troina
- Spain (2):
  - Integrative Pharmacology and Systems Neurosciences, Hospital del Mar Research Institute, Barcelona
  - Servicio de Medicina Interna, Hospital Universitario De La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No